CLINICAL TRIAL: NCT00591526
Title: A Randomized Trial Assessing the Roles of AraC in Newly Diagnosed Acute Promyelocytic Leukemia (APL)
Brief Title: A Randomized Trial Assessing the Roles of AraC in Newly Diagnosed APL Promyelocytic Leukemia (APL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe d'etude et de travail sur les leucemies aigues promyelocytaires (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Centre Hospitalier Universitaire (CHU) of Lille, France., DRC LILLE, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL2000
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Leukemia, Promyelocytic, Acute
Keywords: APL
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (No Intervention): Patients aged ≤ 60 years and with initial WBC ≤ 10000/mm3 Induction treatment
  a) ATRA and chemotherapy ATRA 45 mg/m2/d until hematological CR first intensive chemotherapy course : DNR 60 mg/m2/d during 3 days AraC 200 mg/m2/d during 7 days
  2) Consolidation treatment
  1. First consolidation course (=2nd chemotherapy course) DNR 60 mg/m2/d d1-3 (intravenous bolus injection) AraC 200 mg/m2/d d1-7 (continuous infusion)
  2. Second consolidation course AraC 1g/m2/12h d1-4 (1 hour infusion) Daunorubicin 45 mg/m2/d d1-3 (intravenous bolus injection) 3) Maintenance treatment
  Consists of the combination of continuous low dose chemotherapy and intermittent ATRA, during 2 years
  1. Continuous low dose chemotherapy
  2. Intermittent ATRA
- B (Experimental): Patients aged ≤ 60 years and with initial WBC ≤ 10000/mm3 (Group B) Same treatment as Group A but without AraC.
  Interventions: Drug: Arac
- C (No Intervention): 1. First consolidation course (=2nd chemotherapy course) DNR 60 mg/m2/d d1-3 (intravenous bolus injection) AraC 200 mg/m2/d d1-7 (continuous infusion)
  2. Second consolidation course AraC 1g/m2/12h d1-4 (1 hour infusion) Daunorubicin 45 mg/m2/d d1-3 (intravenous bolus injection)
  CNS prophylaxis : consists of 5 intrathecal (IT) injections of MTX 15mg and AraC 50 mg (12 mg/m2 maximum 15 mg, and 30mg/m2, maximum 50 mg, respectively, in children) + depomedrol IT. I
  3) Maintenance treatment
- D (No Intervention): Patients aged >60 years and initial WBC ≤ 10000/mm3 Induction treatment
  a) ATRA and chemotherapy ATRA 45 mg/m2/d until hematological CR first intensive chemotherapy course : DNR 60 mg/m2/d during 3 days (intravenous bolus injection) NO ARA C DURING THIS FIRST COURSE
  2) Consolidation treatment
  1. First consolidation course DNR 60 mg/m2/d d1-3 AraC 100 mg/m2/d d1-5 G-CSF
  2. Second consolidation course DNR45 mg/m2/d d1-3 AraC 100 mg/m2/d d1-5 G-CSF
     3) maintenance treatment: similar to other groups
  Interventions: Drug: Arac

INTERVENTIONS:
Drug: Arac — Ommit ARAC in the chemotherapy
  Other Names: Cytarabine
  Arms: B; D

SUMMARY:
The first purpose of this randomized trial will be to compare the best treatment group of APL 93 trial (ATRA with early introduction of anthracycline-AraC chemotherapy, followed by 2 consolidation anthracycline-AraC courses and maintenance combining continuous chemotherapy and intermittent ATRA) to the same regimen, but without AraC. It is hoped that the investigational arm, with anthracycline alone chemotherapy (without AraC), will have reduced toxicity without increasing the incidence of relapse, by comparison with a classical induction/consolidation anthracycline-AraC regimen

Thus :

the main end point for this first randomization is relapse at 2 years secondary end points are : complete remission rate ; survival and event free survival at 2 years, and quality-adjusted survival (Q-TWiST).

2) Because patients with initial WBC counts > 10000/mm3 (ie very high counts for APL) appear to remain at relatively high risk of relapse even with the current reference treatment, they will not be included in this trial that assesses the reduction of chemotherapy. On the contrary: i) they will all receive the standard chemotherapy (best treatment group of APL 93 trial);

Thus :

the main end point for this second randomization is relapse at 2 years secondary end points are : survival and event free survival at 2 years 3)Elderly patients with initial WBC ≤ 10000/m3 will receive consolidation chemotherapy without AraC during the first chemotherapy course, and reduced doses of AraC during the second and third course, followed by G-CSF.

DETAILED DESCRIPTION:
All patients will receive induction treatment with ATRA and a first chemotherapy course, followed by two consolidation chemotherapy courses and maintenance with continuous low dose chemotherapy and intermittent ATRA. Initial stratification will be based on age and WBC count.

Patients aged 60 years with initial WBC 10 00 will all receive the reference AraC+ group (Group A ) (no randomization).

Patients with initial WBC > 10000/mm3 will initially all be treated according to the AraC+ group.

Patients > 60 years and with initial WBC ≤ 10000/mm3) will be only registered, without randomization (Group D) and will receive the reference AraC+ group ,but without AraC during the first chemotherapy course ,and with reduced doses of AraC during the second and third course, followed by G-CSF. .

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of APL based on morphological grounds, and which will have to be confirmed by presence of t(15;17) and/or PML-RARα rearrangement (if RT-PCR for APL cannot be performed at your center, send fresh cells to Prof.C.Chomienne, Centre Hayem, Hopital St.Louis, 1 av. Claude Vellefaux, 75475 PARIS or keep frozen RNA [not frozen cells, as the RNA yield for PML-RAR is often poor in those cells]).
* untreated patient
* no contraindication to intensive chemotherapy (especially cardiac contraindication to daunorubicin)
* in female patients : absence of pregnancy and adequate contraceptive method (due to teratogenetic effects of ATRA in early pregnancy)
* written informed consent.

Exclusion Criteria:

* patients already treated
* patients with contraindication to intensive chemotherapy, especially cardiac contraindication to daunorubicin
* in female patients : pregnancy or absence of adequate contraceptive methods

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2000-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
for patients with initial WBC counts > 10000/mm3 - the main end point for this second randomization is relapse at 2 years | 2 years

SECONDARY OUTCOMES:
secondary end points are : complete remission rate ; survival and event free survival at 2 years, and quality-adjusted survival (Q-TWiST). secondary end points are : survival and event free survival at 2 years | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fenaux, MD, Principal Investigator — Assistance Publique Hopitaux de Paris

REFERENCES:
- [Result] Ades L, Chevret S, Raffoux E, de Botton S, Guerci A, Pigneux A, Stoppa AM, Lamy T, Rigal-Huguet F, Vekhoff A, Meyer-Monard S, Maloisel F, Deconinck E, Ferrant A, Thomas X, Fegueux N, Chomienne C, Dombret H, Degos L, Fenaux P; European Acute Promyelocytic Leukemia Group. Is cytarabine useful in the treatment of acute promyelocytic leukemia? Results of a randomized trial from the European Acute Promyelocytic Leukemia Group. J Clin Oncol. 2006 Dec 20;24(36):5703-10. doi: 10.1200/JCO.2006.08.1596. Epub 2006 Nov 20. PMID 17116939